CLINICAL TRIAL: NCT01266304
Title: The Healing Context in CAM: Instrument Development and Initial Validation
Brief Title: The Healing Context in Complementary and Alternative Medicine (CAM): Instrument Development and Initial Validation
Acronym: HEAL
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Carol Greco, Assistant Professor of Psychiatry, University of Pittsburgh
Other Study IDs: AT006453 -1
Record Dates: First submitted 2010-12-16; First posted 2010-12-24 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2015-11

CONDITIONS: Any Condition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- community members: Pittsburgh area community members, including people who attend an integrative medicine clinic and people who attend a conventional medicine clinic.

SUMMARY:
The overall objective of this study is to develop and test an efficient self-report instrument to measure Complementary and Alternative Medicine(CAM)-relevant contextual factors important in healing.

The initial phase of the study involves developing and refining an item bank. During the initial 'item bank development' phase, the investigators will run focus groups and cognitive interviews with individuals who participate in CAM and conventional medicine interventions.

The current protocol in ClinicalTrials.gov pertains only to the initial phase of the study involving focus groups and cognitive interviews.

The next step of instrument development is called Calibration, and will involve administering the revised item bank to an internet sample and to persons who receive services in a CAM clinic and a conventional primary care setting. The items will be calibrated using item response theory and classical test theory. This will result in a computerized adaptive testing version of the instrument, as well as a static short form of the instrument.

The final phase of the project will involve conducting initial validation studies of the instrument. The instrument will be called the Healing Encounters and Attitudes List (HEAL). The investigators will evaluate the convergent, discriminant, and predictive validity of the HEAL in a sample of 200 persons with chronic low back pain who are receiving physical therapy, chiropractic care, or mindfulness-based stress reduction. For convergent validity, the HEAL is expected to display moderate to large correlations with measures of similar constructs. The HEAL is expected to correlate modestly with self-report measures of general psychosocial functioning, in support of discriminant validity. Finally, HEAL score should account for a significant proportion of the variance in treatment outcome, supporting predictive validity.

DETAILED DESCRIPTION:
This project will develop and test a patient self-report measurement tool to assess the perceived contextual factors, such as patient attitudes and expectations, patient provider relationship factors, and environmental factors that contribute to healing. Our project is synergistic with the National Institutes of Health (NIH) Roadmap initiative, Patient Reported Outcomes Measurement Information System (PROMIS), and will use the rigorous instrument development and validation methodology of PROMIS. The overall objective of this study is to develop an efficient self-report instrument to measure CAM-relevant contextual factors important in healing, hereafter referred to as the Healing Encounters and Attitudes List (HEAL), and conduct initial validation in persons seeking CAM and conventional treatment for pain.

Specific Aim 1: Develop an item bank. We will employ several iterative steps used successfully in PROMIS to identify items that assess contextual factors of healing relevant to CAM. Initial steps in developing an item bank include: a) compilation and evaluation of existing instruments and relevant questions, b) consultation with experts, and c) focus groups with individuals who participate in CAM and conventional medicine interventions, and d) item editing. During the initial year of this study, we expect to identify conceptual areas of potential importance to CAM interventions and patients, and identify and edit items to create an item bank assessing these conceptual areas.

Specific Aim 2: Calibrate items. We will use item response theory (IRT) and classical test theory (CTT) to calibrate the items from Aim 1 on three samples: 1) an internet-based sample (n= 1000), 2) 100 outpatients participating in CAM interventions at our Center for Integrative Medicine (CIM), and 3) 100 outpatients at a General Internal Medicine clinic. During year 2-3 we administer the items in the item bank to the 1200 persons, conduct IRT and CTT analyses and refine the item bank to only those items that best assess the constructs. Specific aim 2 will result in a Computerized Adaptive Testing (CAT) version of the HEAL, which maximizes information while minimizing patient time burden. A static short form of the HEAL will be derived from the HEAL CAT in Aim 2.

Specific Aim 3: Conduct initial validation studies. We will evaluate convergent, discriminant, and predictive validity of the Healing Encounters and Attitudes List (HEAL) in a sample of chronic low back pain (CLBP) patients receiving CAM and conventional medicine treatments. The validity studies will use two samples of adults with CLBP: 100 persons receiving CAM treatments: chiropractic manipulation (CM) or mindfulness-based stress reduction (MBSR) at the CIM, and 100 persons receiving conventional care (physical therapy) at Centers for Rehab Services referred by the General Internal Medicine Clinic (GIMC) of the University of Pittsburgh Medical Center (UPMC). We will administer the CAT version of the HEAL questionnaire developed in aims 1 and 2 as well as conventional measures of treatment expectancy, confidence in treatment provider, psychosocial functioning, and treatment outcome measures for CLBP of pain and disability.

* Hypothesis 3a: Scores on the HEAL measure will display moderate to large correlations (r's > .50) with similar self-report measures, supporting convergent validity.
* Hypothesis 3b: Scores on the HEAL measure will correlate modestly (r's = .20-.35) with self-report measures of general psychosocial functioning, supporting discriminant validity.
* Hypothesis 3c: HEAL scores will account for a significant proportion of variance in treatment outcome in both samples. In addition, we predict that HEAL scores will demonstrate incremental validity, i.e., they will account for significant incremental variance in outcome beyond that accounted for by existing measures of treatment expectancy and related constructs.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or over
2. Males and Females
3. able to read, speak and understand English
4. able to complete informed consent procedures

Exclusion Criteria:

1. self reported History of schizophrenia or current psychotic symptoms
2. self reported History of bipolar disorder
3. self report of substance dependence within the past 6 months
4. self reported history of organic neuropsychiatric syndromes (e.g., Alzheimer's, Parkinson's, dementia)
5. Lack of willingness or ability to provide informed consent
6. Subjects may only complete either 1.) focus group or 2.) cognitive interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample, conventional primary care clinic, and integrative medicine clinic.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Transcribed focus group information | Baseline (generally same day as study enrollment, but baseline data collection may occur at a single study visit within 4 weeks of enrollment)
  Participants' opinions regarding factors that contribute to healing, such as important patient characteristics, provider characteristics, and environmental factors.

SECONDARY OUTCOMES:
Cognitive Interviews regarding items | Baseline (generally same day as study enrollment, but data collection may occur at a single study visit within 4 weeks of study enrollment)
  Participants will 'think aloud' while answering items in the HEAL item bank. This will provide the investigative team with information on whether item stems, reponse choices, or wording need to be changed so that they can be easily and accurately understood and answered.

CONTACTS AND LOCATIONS:
Overall Officials: Carol M Greco, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Greco CM, Glick RM, Morone NE, Schneider MJ. Addressing the "It Is Just Placebo" Pitfall in CAM: Methodology of a Project to Develop Patient-Reported Measures of Nonspecific Factors in Healing. Evid Based Complement Alternat Med. 2013;2013:613797. doi: 10.1155/2013/613797. Epub 2013 Dec 19. PMID 24454501
- [Result] Greco CM, Yu L, Johnston KL, Dodds NE, Morone NE, Glick RM, Schneider MJ, Klem ML, McFarland CE, Lawrence S, Colditz J, Maihoefer CC, Jonas WB, Ryan ND, Pilkonis PA. Measuring nonspecific factors in treatment: item banks that assess the healthcare experience and attitudes from the patient's perspective. Qual Life Res. 2016 Jul;25(7):1625-34. doi: 10.1007/s11136-015-1178-1. Epub 2015 Nov 12. PMID 26563249
- See also: PROMIS network website — http://www.nihpromis.org